CLINICAL TRIAL: NCT01332344
Title: Comparison of Healthcare Utilization and Costs in Patients With Asthma Who Fluticasone/Salmeterol Inhalation Powder Versus Other Inhaled Corticosteroid(s) in Typical Clinical Practice Using Health Insurance Claims Data.
Brief Title: Outcomes in Patients Taking Fluticasone Propionate/Salmeterol Combination or Other Inhaled Corticosteroids
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112604
Record Dates: First submitted 2010-03-04; First posted 2011-04-11 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: fluticasone propionate/salmeterol combination; Asthma; inhaled corticosteroids; outcomes
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma patients treated with inhaled corticosteroids: Asthma subjects newly prescribed inhaled corticosteriods
  Interventions: Drug: Fluticasone propionate/salmeterol combination; Drug: Inhaled corticosteroids

INTERVENTIONS:
Drug: Fluticasone propionate/salmeterol combination — Asthma subjects newly prescribed fluticasone propionate/salmeterol combination
Drug: Inhaled corticosteroids — asthma subjects newly prescribed inhaled corticosteroids in clinical practice

SUMMARY:
The objective of this study is to compare healthcare utilization and costs in asthma patients who receive fluticasone propionate/salmeterol combination 100mcg/50mcg ("FSC 100/50") or inhaled corticosteriods in typical clinical practice using a retrospective observational cohort study design of large managed care database.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with asthma as determined by ICD-9 codes and asthma drug use
* at least 12 years of age
* treated with inhaled corticosteroids

Exclusion Criteria:

* Subjects with COPD or treatment for COPD

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study intends to identify subjects with asthma treated with inhaled corticosteroids
Sampling Method: Probability Sample
Enrollment: 5180 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To assess the difference in asthma related exacerbations | 90 days post index
  Asthma related exaceberation is defined as any asthma related emergency department visit, or inpatient visit or oral corticosteroid dispensing.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline